CLINICAL TRIAL: NCT01327417
Title: Cortical/Subcortical Circuits in Late-Life Depression
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2009-0613; R01MH073989 (NIH)
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Depression
Keywords: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Depressed: Patients with Major Depressive Disorder
- Healthy Controls

SUMMARY:
The purpose of the study is to examine the relationship between brain structure and depression in adults aged 60 or older. This relationship is determined using magnetic resonance imaging technology (MRI), a scanner with a magnet that is used to create images of the brain.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) and other clinically significant forms of "minor depression" are among the most common mental disorders in the elderly. Data from the Epidemiologic Catchment Area Studies indicate that in the community dwelling elderly, the prevalence of MDD is approximately 1-2 percent. The prevalence of dysthymia and "clinically significant" depressive symptoms is estimated to be 2-3% and 5-10% respectively. Clinically significant mood disorders are responsible for considerable medical and psychosocial morbidity. These include frequent medical and psychiatric hospitalizations, visits to the emergency room, suicide attempts, and use of alcohol, and other prescription medications with psychotropic effects. The clinical impact of these disorders is comparable to those caused by other chronic medical disorders.

The vast majority of patients with mood disorders are managed at ambulatory care/primary care settings around the country. Ambulatory care clinics have become "defacto" settings for the diagnosis and management of psychiatric problems, especially in the elderly. Depression, particularly in the elderly, is associated with several chronic medical illnesses including malignancies, chronic obstructive pulmonary disease, and gastrointestinal, vascular, autoimmune and demyelinating disorders. Acknowledging the overall robust association between medical illness and mood disorders, the NIH consensus statement on depression in the elderly states, "The hallmark of depression in late-life is its association with medical comorbidity." While the precise mechanisms by which coexisting medical illnesses contribute to depression remain unclear, neuroanatomical, vascular, immunologic, psychosocial and /or a combination of these mechanisms have been invoked as possible pathways by which medical disorders may lead to depression in the elderly.

Late-life MDD is characterized by 1) Neuroanatomical changes in neocortical and subcortical regions of the brain. These principally comprise a decrease in focal brain volumes and an increase in the volume of high intensity lesions in the parenchyma; 2) The increase in high intensity lesions occurs largely, though not exclusively, in the white matter; 3) Preliminary studies suggest that there are abnormalities in white matter regions and tracts even in areas that appear normal in MR images in patients with late-life MDD when compared with controls; 4) Biochemical and biophysical changes in the white matter are likely related to the pathophysiology of major psychiatric disorders independent of the impact of cerebrovascular disease/risk factors.

TRIAL OBJECTIVES AND PURPOSE

Specific Aim 1: To estimate absolute levels and ratios (metabolite/creatine) of NAA, Ch and Ml bilaterally in the dorsolateral white matter and subcortical nuclei in patients with MDD and non-depressed controls.

Hypothesis: Absolute levels and ratios of Ch and Ml will be higher and levels of NAA will be lower in the dorsolateral white matter and the subcortical nuclei in patients with MDD when compared with controls.

Specific Aim 2: To estimate magnetization transfer ratios (MTR) bilaterally in the frontal white matter/head of the caudate nucleus and the putamen in patients with MDD and controls and to examine the relationship between MTR and MRS measures in the dorsolateral white matter. Hypothesis a: MTR will be significantly lower in normal appearing dorsolateral white matter regions and subcortical nuclei (caudate nucleus and putamen) in patients with MDD when compared with controls.

Hypothesis b: There will be an inverse relationship between MTR and normalized levels of Ml in patients diagnosed with MDD in the dorsolateral white matter bilaterally.

Specific Aim 3: To examine the neurocognitive correlates of frontal and striatal compromise identified using MRS and MT ratio measures in patients with MDD and controls. The associations between NAA and a global cognitive scale and MT ratios from the bilateral dorsolateral white matter and subcortical nuclei and subscales targeted to dorsolateral and striatal cognitive functioning will be examined.

Hypothesis a: Among healthy and depressed elderly, NAA/Cr with be positively related to a global scale of cognitive function.

Hypothesis b: Among healthy and depressed elderly, MT ratios of the dorsolateral cortices will be positively related to a subscale of dorsolateral function (working memory, executive function, nonverbal recall).

Hypothesis c: Among healthy and depressed elderly, MT ratios of subcortical nuclei will be positively related to a subscale of striatal function (processing, learning).

Exploratory analyses: In addition to the specific aims above, the investigators will conduct two three exploratory analyses.

Analysis 1: A more finely grained analysis in which the investigators examine the relationship of NAA, Ml and Cho ratios to dorsolateral and striatal subscales after examining their relationship to global cognitive function. The investigators will also study the relationship of the relative concentrations of NAA to Ml (NAA/MI) and Ch (NAA/Ch) to global and regional subscales. In addition, the preliminary MTR data suggest that there may be laterally effects, which the investigators will examine.

Analysis 2: A comparison of blood samples of the healthy versus depressed subject groups, to see if there is evidence of differences in the neurotransmitter system, hypothalamic-pituitary-adrenals (HAP) axis, and immune function between these two groups of elderly persons.

Analysis 3: To examine whether neuroimaging and cognitive measures associated with major depression are reversed by antidepressant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 60 years or greater
* Diagnosis of major depressive disorder using standard diagnostic and statistical manual (DSM) criteria
* Score of 15 or greater on the 17-item Hamilton Depression rating scale
* Mini Mental Status Exam score of 24 or greater
* No evidence of clinical dementia or any other clinical brain disorder
* Free of psychotropic/psychoactive medications for at least 2 weeks

Exclusion Criteria:

* Presence of dementia or any other clinical brain disorder (Parkinson's, Alzheimer's)
* History of progressive cognitive decline and/or Mini Mental Status Exam score of less than 24
* Lifetime diagnosis of substance abuse
* Unstable medical illness (grade 4 on the Cumulative Illness Rating Scale)
* Presence of any metallic implant that would preclude an MRI scan (pacemaker, etc.)
* Concurrent Axis 1 disorder (schizophrenia, bipolar)
* Psychotropic medication implicated in depression i.e. Reserpine, Alpha methyl dopa, Beta blockers, multiple long acting benzodiazepines (valium, flurazepam, chlordiazepoxide), neuroleptics;
* Seizure disorder
* Stroke/Transient Ischemic Attack
* Central nervous system disorder (Parkinson's disease, multiple sclerosis)
* Trauma to head/Loss of Consciousness
* Claustrophobia
* Eating disorder (anorexia, bulimia)
* Weight of over 350 pounds
* Learning disorder (dyslexia, ADHD)
* Psychosis, panic or anxiety disorder outside the context of depression
* Mood stabilizing agents such as lithium and Divalproex sodium and antidepressants - as they have been shown to impact on brain levels of NAA, Ch and Ml

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Geriatric Medicine and Psychiatry clinics within the UIC Medical Center. Patients with mood and other psychiatric disturbances are frequently referred by physicians from both geriatric medicine and family medicine for a consultation and sometimes for ongoing psychiatric care.
  * Community outreach efforts and recruitment through advertising in newsletters, local newspapers
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2009-09-22 (Actual); Primary Completion 2014-08-19 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anand Kumar, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois, Chicago, Illinois, United States

REFERENCES:
- [Background] Ballmaier M, Narr KL, Toga AW, Elderkin-Thompson V, Thompson PM, Hamilton L, Haroon E, Pham D, Heinz A, Kumar A. Hippocampal morphology and distinguishing late-onset from early-onset elderly depression. Am J Psychiatry. 2008 Feb;165(2):229-37. doi: 10.1176/appi.ajp.2007.07030506. Epub 2007 Nov 6. PMID 17986679
- [Background] Ballmaier M, Kumar A, Elderkin-Thompson V, Narr KL, Luders E, Thompson PM, Hojatkashani C, Pham D, Heinz A, Toga AW. Mapping callosal morphology in early- and late-onset elderly depression: an index of distinct changes in cortical connectivity. Neuropsychopharmacology. 2008 Jun;33(7):1528-36. doi: 10.1038/sj.npp.1301538. Epub 2007 Aug 22. PMID 17712348
- [Background] Lavretsky H, Ballmaier M, Pham D, Toga A, Kumar A. Neuroanatomical characteristics of geriatric apathy and depression: a magnetic resonance imaging study. Am J Geriatr Psychiatry. 2007 May;15(5):386-94. doi: 10.1097/JGP.0b013e3180325a16. PMID 17463189
- [Result] Kumar A, Ajilore O. Magnetic resonance imaging and late-life depression: potential biomarkers in the era of personalized medicine. Am J Psychiatry. 2008 Feb;165(2):166-8. doi: 10.1176/appi.ajp.2007.07111771. No abstract available. PMID 18245182
- See also: Related Info — http://www.psych.uic.edu/